CLINICAL TRIAL: NCT01075204
Title: Clarithromycin Modified Release Observational Study for Evaluation of Treatment, Tolerability & Recovery Time in Saudi & Egyptian Clinical Settings (CLOSER)
Acronym: CLOSER
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Eilaf (Other)
Responsible Party: Sponsor
Other Study IDs: P11-989
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory Tract Infection; Clarithromycin; Recovery
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clarithromycin modified release: Patients with upper or lower respiratory tract infection were administered clarithromycin modified release 500 mg once daily for 7 days and then followed for a further 3 days, per routine clinical practice.
  Interventions: Drug: clarithromycin modified release 500 mg

INTERVENTIONS:
Drug: clarithromycin modified release 500 mg — clarithromycin modified release 500 mg for 7 days
  Other Names: Clarithromycin Modified Release 500 mg (Klacid XL)

SUMMARY:
The objective is to describe the time to recovery of symptoms (cough, mucus, fever, sore throat, and others), tolerability and compliance of treatment with clarithromycin once daily in patients with upper or lower respiratory tract infections in the routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults, equal to or more than 18 years years of age
* Patients with respiratory tract infections, including any of the following:

  * Acute tracheitis, acute tracheobronchitis
  * Acute sinusitis
  * Chronic sinusitis
  * Acute tonsillopharyngitis
  * Acute bronchitis
  * Mild community-acquired pneumonia
  * Acute exacerbation of chronic bronchitis

Exclusion Criteria:

* Known hypersensitivity to or previously intolerant of macrolides.
* Illness severe enough to warrant hospitalization or parenteral therapy.
* Concomitant use of any of the following medications:

  * Drugs metabolized by CYP3A isozyme: alprazolam, astemizole, carbamazepine, cilostazol, cisapride, cyclosporin, disopyramide, ergot alkaloids, lovastatin, methylprednisolone, midazolam, omeprazole, oral anticoagulants (e.g. warfarin), pimozide, quinidine, rifabutin, sildenafil, simvastatin, tacrolimus, terfenadine, triazolam and vinblastine.
  * Drugs metabolized by other isozymes within CYP450 system: phenytoin, theophylline and valproate.
  * Colchicine, Digoxin, Some antiretrovirals: zidovudine and ritonavir.
* Severe immunodeficiency and chronic disease conditions.
* Renal or hepatic impairment (creatinine clearance under 30 mL/min, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and gamma-glutamyltransferase (GGT) equal or more than 3x higher level in comparison with the norm).
* Mental condition rendering the subject unable to understand the nature of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assignment to clarithromycin therapy falls within current clinical practice and was not decided in advance by this protocol. Study participants were selected from patients seen at the primary care clinic, with a preliminary clinical diagnosis of an upper or lower respiratory tract infection who were considered for antibiotic treatment and prescribed clarithromycin.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tahoun, Bachelor, Study Director — Abbott Laboratories - Saudi Arabia
Locations (12):
- Egypt (11):
  - Site Ref # / Investigator 50162, Cairo
  - Site Ref # / Investigator 50215, Cairo
  - Site Ref # / Investigator 50225, Cairo
  - Site Ref # / Investigator 50235, Cairo
  - Site Ref # / Investigator 50236, Cairo
  - Site Ref # / Investigator 50237, Cairo
  - Site Ref # / Investigator 51204, Cairo
  - Site Ref # / Investigator 51205, Cairo
  - Site Ref # / Investigator 50213, Helwan
  - Site Ref # / Investigator 51206, Tanta
  - Site Ref # / Investigator 51207, Tanta
- Site Ref # / Investigator 22543, Jeddah, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Groups:
- Clarithromycin Modified Release: Participants with upper or lower respiratory tract infection were administered clarithromycin modified release 500 mg once daily for 7 days and then followed for a further 3 days, per routine clinical practice.
Period: Overall Study
Arm/Group | Clarithromycin Modified Release
Started | 335
Completed | 335
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
Age Continuous [Mean (Standard Deviation); unit: years] — Age data provided for 330 participants.
  years | 35.48 (12.552)
Sex/Gender, Customized [Number; unit: participants]
  Male | 205
  Female | 122
  Missing | 8
Region of Enrollment [Number; unit: participants]
  Egypt | 120
  Saudi Arabia | 215

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Fast Recovery
Description: Fast recovery is defined as the resolution of symptoms within 5 days or less from the start of clarithromycin modified release treatment. Recovery is defined as returning to the symptom status prior to the onset of the respiratory tract infection, based on the participant and physician's assessment.
  Data are reported for all symptoms taken together (all symptoms resolved within 5 days) and for each individual symptom.
Time Frame: Day 1 to Day 5
Population: All enrolled participants. For the individual symptoms, N indicates the number of participants with that symptom at Baseline and with available recovery data.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
percentage of participants
  All symptoms together [N=335] | 12.8
  Fever response [N=184] | 54.3
  Cough response [N=215] | 27.4
  Sputum response [N=212] | 29.7
  Dyspnea response [N=62] | 37.1
  Abnormal breath sounds response [N=47] | 42.6
  Rhinorrhea response [N=113] | 28.3
  Nasal congestion response [N=233] | 33.5
  Post-nasal discharge response [N=178] | 18.5
  Sneezing response [N=87] | 25.3
  Sore throat response [N=200] | 38.0
  Painful swallowing response [N=162] | 38.9
  Itchy watery eye response [N=33] | 6.1
  Malaise response [N=68] | 30.9
  Myalgia response [N=79] | 34.2

2. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure is defined as failure to return to baseline symptom status (symptom status prior to the onset of the respiratory tract infection) within 10 days or the need for new treatments or medications during the first 10 days for persistence or aggravation of symptoms.
  Participants with treatment failure were further categorized as:
  * All symptoms improved but not resolved within the study period;
  * Some symptoms improved and some resolved;
  * Some symptoms resolved or improved while other symptoms did not improve (unchanged);
  * Some symptoms resolved or improved while other symptoms became worse.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
percentage of participants
  Treatment failure total | 13.1
  All symptoms improved but not resolved | 0.9
  Some symptoms improved and some resolved | 3.9
  Some symptoms resolved/improved, others unchanged | 6.9
  Some symptoms resolved/improved/others worsened | 1.5

3. Secondary Outcome: Factors Affecting the Speed of Recovery
Description: Factors affecting the speed of recovery were examined and tested for association with the speed of recovery. Logistic regression was conducted to assess whether the following nine variables; age, gender, body mass index (BMI), concomitant tobacco use, steroid use, bronchial asthma, allergic rhinitis, nasal septum deviation and chronic obstructive pulmonary disease (COPD) act as predictors for speed of recovery of respiratory tract infections. Data shown are the beta regression coefficients for each variable.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: coefficient
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
coefficient
  Age | -0.007
  Gender | 0.216
  Body mass index (BMI) | 0.004
  Tobacco use | 0.419
  Steroid use | -0.456
  Bronchial asthma | 0.140
  Allergic rhinitis | 19.292
  Nasal septum deviation | 18.698
  Chronic obstructive pulmonary disease (COPD) | 19.281
Statistical Analysis 1: Comparison: Clarithromycin Modified Release; Logistic regression: Omnibus Test of Model Coefficients (all the nine variables are considered together); Test type: Superiority or Other; p = 0.334, Chi-squared; 9 degrees of freedom

4. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient, which does not necessarily have a causal relationship with their treatment.
  If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE):
  Results in death or is life-threatening, results in admission or prolongation of hospitalization, is a congenital anomaly or persistent or significant disability/incapacity or is an important medical event requiring medical or surgical intervention to prevent any of the outcomes listed above.
  Please see Adverse Events section below for more details.
Time Frame: 10 days
Population: All enrolled patients.
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Any adverse event | 2
  Serious adverse event | 0

5. Primary Outcome: Percentage of Participants With Clinical Success
Description: Clinical success is defined as the disappearance of cough and other symptoms within 10 days or less from the start of clarithromycin treatment.
Time Frame: 10 days
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
percentage of participants | 86.9 [83.28 to 90.52]

6. Primary Outcome: Classification of Overall Response
Description: Based on the participant and physician's assessment, overall symptom response was classified as follows:
  * Fast Responders: participants showing clinical recovery of all symptoms within the first 5 days of treatment.
  * Slow Responders: participants showing clinical recovery between Day 6 & Day 10 (includes participants with a fast response for some symptoms and slow response for the remaining symptoms).
  * Failure response: participants showing no clinical success by Day 10, or showing need for another anti-infective treatment to resolve aggravated symptoms (includes participants with a failure response for some symptoms and either a slow or fast response for the remaining symptoms).
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Fast responders | 43
  Slow responders | 248
  Failure response | 44

7. Secondary Outcome: Fever Status at End of Study
Description: Participants with fever (temperature over 37.0 degree of Celsius) at any time during the study were classified at the end of study as resolved, improved or no change. 'No fever' indicates participants with no fever during the study period.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Resolved | 120
  Improved | 70
  No change | 5
  No fever | 140

8. Secondary Outcome: Cough Status at End of Study
Description: Participants with cough at any time during the study were classified at the end of study as resolved, improved, became worse, or no change. 'No cough' indicates participants with no cough symptoms during the study period.
Time Frame: 10 days
Population: Enrolled patients with cough data available.
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 333
participants
  Resolved | 93
  Improved | 100
  No change | 23
  Worsened | 4
  No cough | 113

9. Secondary Outcome: Sputum Status at End of Study
Description: Participants with sputum symptoms at any time during the study were classified at the end of study as resolved, improved, became worse, or no change. 'No sputum' indicates participants with no sputum symptoms during the study period.
Time Frame: 10 days
Population: Enrolled patients with sputum data available.
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 333
participants
  Resolved | 88
  Improved | 102
  No change | 19
  Worsened | 4
  No sputum | 120

10. Secondary Outcome: Dyspnea Status at End of Study
Description: Participants with dyspnea (shortness of breath) at any time during the study were classified at the end of study as resolved, improved, became worse, or no change. 'No dyspnea' indicates participants with no dyspnea symptoms during the study period.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Resolved | 31
  Improved | 28
  No change | 2
  Worsened | 1
  No dyspnea | 273

11. Secondary Outcome: Abnormal Breathing Sounds Status at End of Study
Description: Participants with abnormal breathing sounds such as wheezing or rales at any time during the study were classified at the end of study as resolved, improved, or no change. 'No abnormal breath sounds' indicates participants with no abnormal breathing sounds during the study period.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Resolved | 30
  Improved | 13
  No change | 4
  No abnormal breath sounds | 288

12. Secondary Outcome: Rhinorrhea Status at End of Study
Description: Participants with rhinorrhea (runny nose) at any time during the study were classified at the end of study as resolved, or no change. 'No rhinorrhea' indicates participants with no rhinorrhea during the study period.
Time Frame: 10 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
participants
  Resolved | 55
  Improved | 56
  No change | 2
  No rhinorrhea | 222

13. Secondary Outcome: Post-nasal Discharge Status at End of Study
Description: Participants with post-nasal discharge at any time during the study were classified at the end of study as resolved, improved, or no change. 'No post-nasal discharge' indicates participants with no post-nasal discharge symptoms during the study period.
Time Frame: 10 days
Population: Enrolled patients with post-nasal discharge data available.
Measure: Number; unit: participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 333
participants
  Resolved | 75
  Improved | 98
  No change | 6
  No post-nasal discharge | 154

14. Secondary Outcome: Percentage of Participants Compliant With Treatment
Description: Treatment compliance was assessed by the study physician at each study visit. The percentage of participants who were compliant with study treatment for 6 days, 7 days and 8 days is reported.
Time Frame: 10 days
Population: All enrolled patients.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin Modified Release
Number analyzed (Participants) | 335
percentage of participants
  6 days | 43
  7 days | 54
  8 days | 3

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Clarithromycin Modified Release
Serious Adverse Events (participants affected / at risk) | 0/335
Other Adverse Events (participants affected / at risk) | 2/335
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clarithromycin Modified Release (N=335)
Dyspepsia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.